CLINICAL TRIAL: NCT05067218
Title: Effect of External Cold and Vibration (Buzzy Device) Versus the Conventional Technique on Pain Perception During Local Anesthesia Injection in Children.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mai Gamal Eldeen Hassan Sabra, principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Buzzy device in Children.
Record Dates: First submitted 2021-09-22; First posted 2021-10-05 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Anesthesia; Anesthesia, Local; Vibration

STUDY DESIGN:
Intervention Model Description: split mouth
Who Masked: Outcomes Assessor
Masking Description: Blinding of the operator and the patients will not be applicable due to the difference between the used techniques, however, the statistician will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- buzzy device (intervention) (Active Comparator): The wings of buzzy device will be kept frozen and once the child is ready, the frozen wing will be attached to the device and Buzzy will be placed extra-orally above the area/cheek where local anesthetic is to be delivered.
  Interventions: Device: buzzy device
- Conventinal anasthesia ( control ) (Experimental): * The site of injection will be dried then topical anesthetic gel of 20% benzocaine (Dharma Ophal-S) will be applied. The duration of application of gel will be 1 minute.
  * Local anesthetic solution will be delivered using a standard aspirating syringe with 27-gauge, 21 mm short needles.
  Interventions: Other: Conventinal anasthesia

INTERVENTIONS:
Device: buzzy device — bee shaped with wings could be frozen.
  Arms: buzzy device (intervention)
Other: Conventinal anasthesia — normal technique of injection
  Arms: Conventinal anasthesia ( control )

SUMMARY:
This study adopts the null hypothesis (There is no difference in pain perception during local anesthesia injection with the buzzy device in comparison to the conventional technique).

DETAILED DESCRIPTION:
The injection of local anesthesia in children is usually associated with fear, anxiety, and discomfort. There is an essential need to develop techniques that decrease pain during injection, preventing patients from avoiding dental treatment.The efficacy of a child-friendly device, having a combined effect of vibration and distraction, with the conventional method of injection on pain, anxiety, and behavior of pediatric patients. The evaluation the pain perception and comfort of the patient during local anesthesia delivery using the Buzzy device and conventional syringe and revealed that the external cold and vibration via Buzzy can reduce pain and anxiety during local anesthetic delivery for various dental procedures.

ELIGIBILITY:
Inclusion Criteria:

* Children classified as cooperative or potentially cooperative according to Wright's classification of child behaviour.
* Medically fit children (ASA I, II).
* Children mentally capable of communication.
* Children aged 6-11 years.
* First dental visit.
* Patient requiring inferior alveolar nerve block local anesthesia injection for dental treatment.

Exclusion Criteria:

* Children with a behavioral management problem.
* Children with known allergy to local anesthetic agents.
* Parental refusal for participation

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 12 (Estimated)
Dates: Start 2021-10-15 (Estimated); Primary Completion 2022-10-15 (Estimated); Study Completion 2022-11-15 (Estimated)

PRIMARY OUTCOMES:
Pain perception during LA injection | one hour
  by wong baker scale

SECONDARY OUTCOMES:
Heart rate during injection of local anesthesia. | one hour
  pulse oximeter

OTHER OUTCOMES:
Child's behavior during local anesthesia injection. | one hour
  FLACC scale